CLINICAL TRIAL: NCT03928782
Title: Study on Dose-effect Relationship Between Radiation Injury Dose and Expression of Associated microRNAs in Human Peripheral Blood
Brief Title: Dose-effect Relationship Between microRNAs in Peripheral Blood and Radiation Injury
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Affiliated Hospital to Academy of Military Medical Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: KY-2018-4-26
Record Dates: First submitted 2019-04-24; First posted 2019-04-26 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Radiation Injuries, Experimental
Keywords: Radiation Injuries; microRNA
MeSH Terms: conditions — Radiation Injuries, Experimental; Radiation Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: 5 Gy or 10 Gy units of whole-body radiation — 8 subjects will be received 5 Gy units of whole-body radiation or 10 Gy units of whole-body radiation.

SUMMARY:
Rapid and accurate assessment of radiation injury dose is the key to success in early treatment and an urgent issue to be solved in clinical medicine.Researches showed that the expression of the microRNAs in human peripheral blood had much correlation with radiation injury resulted from different dosages of radiation.In this study,acute leukemic patients who will be pretreated by whole-body radiation are taked as the object of study,and biochip technology are adopted to detect the expression levels of the microRNAs in subject peripheral blood before-and-after radiation,and different expression is tested and Bioinformatics prediction,to evaluate the correlation between radiation injury dose and expression levels of the microRNAs in human peripheral blood.

ELIGIBILITY:
Inclusion Criteria:

* subjects who suffer from acute leukemic subjects who accept chemotherapy within one month and will be pretreated by whole-body irradiation peripheral blood cells of subjects are approximate to those of healthy person aged between 18 and 50 years old subjects who are competent to give written informed consent subjects without other systemic diseases

Exclusion Criteria:

* subjects who suffer from serious other systemic diseases subjects who are unwilling or unable to cooperate with this clinical study other serious cases that probably hinder this clinical study

Ages: 18 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: Acute leukemic patients after chemotherapy,who will be pretreated by whole-body irradiation
Sampling Method: Non-Probability Sample
Enrollment: 8 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-07-01 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
expression levels of the microRNAs | 12 hours
  the expression levels of the microRNAs in human peripheral blood before radiation，12 hours after radiation and 24 hours after radiation

CONTACTS AND LOCATIONS:
Overall Officials: Lu rongjian, doctor, Study Chair — Chinese PLA 307 Hospital; Guo biao, master, Study Director — Chinese PLA 307 Hospital
Locations (1):
- Chiese PLA 307 hospital, Beijing, Beijing Municipality, China